CLINICAL TRIAL: NCT00334594
Title: Neoadjuvant Chemotherapy and Extrapleural Pneumonectomy of Malignant Pleural Mesothelioma (MPM) With or Without Hemithoracic Radiotherapy. A Randomized Multicenter Phase II Trial
Brief Title: Pemetrexed Disodium and Cisplatin Followed by Surgery With or Without Radiation Therapy in Treating Patients With Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 17/04; SWS-SAKK-17/04; EU-20615; 2006-000445-19 (EudraCT Number); LILLY-SAKK-17/04 (Other: SAKK); CDR0000481153
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Malignant Mesothelioma
Keywords: epithelial mesothelioma; sarcomatous mesothelioma; stage IA malignant mesothelioma; stage IB malignant mesothelioma; stage II malignant mesothelioma; stage III malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Solitary Fibrous Tumor, Pleural | interventions — Cisplatin; Pemetrexed; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No radiotherapy (Active Comparator)
  Interventions: Drug: Cisplatin; Drug: Pemetrexed; Procedure: Therapeutic conventional surgery
- Radiotherapy (Experimental)
  Interventions: Drug: Cisplatin; Drug: Pemetrexed; Procedure: Therapeutic conventional surgery; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 75 mg/m2 i.v. over approximately 2 hours on day 1 every 21 days
Drug: Pemetrexed — Pemetrexed 500 mg/m2 i.v. over approximately 10 minutes on day 1 every 21 days
Procedure: Therapeutic conventional surgery — Extrapleural pneumonectomy
Radiation: Radiotherapy — CTV1 will receive 45 or 46 Gy. CTV2 will be treated up to a total dose of 55,9 to 56,2 Gy.
  Arms: Radiotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as pemetrexed disodium and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation therapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This randomized phase II trial is studying how well giving pemetrexed disodium together with cisplatin followed by surgery with or without radiation therapy works in treating patients with malignant pleural mesothelioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the short-term outcomes and feasibility of neoadjuvant therapy with pemetrexed disodium and cisplatin followed by extrapleural pneumonectomy in patients with malignant pleural mesothelioma.
* Evaluate the long-term outcomes and feasibility of postoperative hemithoracic radiotherapy in patients with R0 or R1 resection.

Secondary

* Determine the quality of life of these patients.
* Identify predictive and prognostic markers in these patients.
* Determine relapse-free or progression-free survival and overall survival of these patients.
* Collect tissue and blood from these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, histology (sarcomatous or other vs epithelial or mixed histology), nodal status (N0-1 vs N2), and extent of disease (T1-2 vs T3).

* Part 1 (neoadjuvant therapy and surgery): Patients receive pemetrexed disodium IV over 10 minutes and cisplatin IV over 2 hours on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Within 8 weeks after completion of neoadjuvant therapy, patients without progressive disease undergo extrapleural pneumonectomy.
* Part 2 : Patients achieving R0 or R1 resection proceed to part 2 of study treatment and are randomized to 1 of 2 treatment arms. Patients with R2 resection, disease progression, or symptomatic deterioration after treatment in part 1 are taken off study.

  * Arm I (no postoperative radiotherapy): Patients do not undergo radiotherapy. Quality of life is assessed at baseline and at 6, 10, 16, and 22 weeks after randomization.
  * Arm II (postoperative radiotherapy): Beginning within 10 weeks after surgery, patients undergo radiotherapy to the hemithoracic region 5 days a week for approximately 5 weeks in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at baseline and at 4, 8, 14, and 20 weeks after initiation of radiotherapy.

Patients undergo blood and tissue collection at registration and surgery for laboratory and biomarker analysis.

After completion of study treatment, patients are followed periodically for up to 5 years after surgery.

PROJECTED ACCRUAL: A total of 155 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed malignant pleural mesothelioma

  * T1-3, N0-2, M0 disease according to International Mesothelioma Interest Group staging system
* No obvious invasion of mediastinal structures by CT scan (e.g., heart, aorta, spine, esophagus)
* No obvious widespread chest wall invasion

  * Resectable chest wall lesions allowed

PATIENT CHARACTERISTICS:

* WHO performance score 0-1
* Fit for neoadjuvant therapy, surgery, and postoperative radiotherapy
* Creatinine clearance > 60 mL/min
* Hemoglobin ≥ 10.0 g/dL
* WBC ≥ 3,500/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 1.5 times ULN
* Alkaline phosphatase ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for up to 12 months after completion of study treatment
* FEV_1 ≥ 40% of predicted based on spirometry and lung perfusion scan, if necessary
* No serious underlying medical condition that would preclude study requirements (e.g., active autoimmune disease or uncontrolled diabetes)
* No known hypersensitivity against pemetrexed disodium, cisplatin, or other platinum-containing substances or any other components used for the preparation of the drugs
* No restricted power of hearing (especially in the upper frequency range)
* No acute infections

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy
* No treatment on another clinical trial within the past 30 days
* No prior pleurectomy or lung resection
* No prior radiotherapy of the lower neck, thorax, or upper abdomen
* No aspirin, cyclooxygenase-2 inhibitors, or nonsteroidal anti-inflammatory agents for 5 days prior to, during, and for 2 days after pemetrexed disodium administration
* No other concurrent experimental drugs or anticancer therapy
* No concurrent drugs that would contraindicate study drugs
* No concurrent vaccination against yellow fever

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2005-11-14 (Actual); Primary Completion 2014-03-26 (Actual); Study Completion 2018-01-23 (Actual)

PRIMARY OUTCOMES:
Complete macroscopic resection (part 1) | After surgery (15 weeks after trial registration)
Loco-regional relapse-free survival (part 2) | From surgery until the first occurrence of loco-regional relapse

SECONDARY OUTCOMES:
Response to neoadjuvant therapy (part 1) | Every 6 months in the follow-up until death for a maximum of 5 years
Adverse drug reaction to neoadjuvant therapy (part 1) | According to CTCAE
Operability (part 1) | Proportion of patients remaining operable after completing chemotherapy (9 weeks after trial registration)
Surgical complications (part 1) | Within 3 month after surgery
Reasons for non-randomization (part 1) | Reasons for non-randomization include macroscopic incomplete resection, patients' refusal or patient can not be subjected to RT within 10 weeks after surgery.
Relapse-free or progression-free survival (part 1) | From registration until progression/relapse (loco-regional or distant) or death
Adverse reaction to postoperative radiotherapy (part 2) | According to CTCAE
Late toxicity (part 2) | Late toxicities occurring later than 6 weeks after the last RT fraction
Feasibility of postoperative radiotherapy (part 2) | Proportion of patients receiving at least 90% of planned RT dose
Relapse-free survival (part 2) | From registration until progression/relapse (loco-regional or distant) or death
Psychological distress (quality of life) (part 2) | Until 22 weeks after treatment termination
Overall survival | From registration until death for all registered patients, and from randomization to death for all randomized patients.

CONTACTS AND LOCATIONS:
Overall Officials: Rolf A. Stahel, Prof, Study Chair — UniversitaetsSpital Zuerich
Locations (13):
- Universitaetsklinikum Freiburg, Freiburg im Breisgau, Germany
- Switzerland (12):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitaetsspital-Basel, Basel
  - Spital Tiefenau, Bern
  - Inselspital Bern, Bern
  - Kantonsspital Bruderholz, Bruderholz
  - Kantonsspital Graubuenden, Chur
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Olten, Olten
  - Kantonsspital - St. Gallen, Sankt Gallen
  - SpitalSTS AG Simmental-Thun-Saanenland, Thun
  - UniversitaetsSpital Zuerich, Zurich

REFERENCES:
- [Result] Stahel RA, Riesterer O, Xyrafas A, Opitz I, Beyeler M, Ochsenbein A, Fruh M, Cathomas R, Nackaerts K, Peters S, Mamot C, Zippelius A, Mordasini C, Caspar CB, Eckhardt K, Schmid RA, Aebersold DM, Gautschi O, Nagel W, Topfer M, Krayenbuehl J, Ribi K, Ciernik IF, Weder W. Neoadjuvant chemotherapy and extrapleural pneumonectomy of malignant pleural mesothelioma with or without hemithoracic radiotherapy (SAKK 17/04): a randomised, international, multicentre phase 2 trial. Lancet Oncol. 2015 Dec;16(16):1651-8. doi: 10.1016/S1470-2045(15)00208-9. Epub 2015 Nov 2. PMID 26538423